CLINICAL TRIAL: NCT01677611
Title: Effects of Resveratrol in Patients With Type 2 Diabetes: The RED Trial
Brief Title: Effects of Resveratrol in Patients With Type 2 Diabetes
Acronym: RED
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Khoo Teck Puat Hospital (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Principal Investigator, Kian Peng Goh, Consultant, Khoo Teck Puat Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NIG 35
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Type 2 Diabetes
Keywords: Resveratrol; SIRT1; AMPK
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resveratrol (Experimental): Trans-resveratrol extract from Polygonum Cuspidatum (Mega Resveratrol, Danbury, USA) was used in the trial.Following the run-in period, subjects who were tolerant of the placebo would proceed to the treatment period. Subjects were given a starting dose of 500 mg daily of either resveratrol.The dose was increased by 500 mg per day every 3 days to a maximum dose of 3 g per day in three divided doses if there was no hypoglycemia. Subjects were instructed to abstain from foods with high resveratrol content during the entire duration of the trial.
  Interventions: Drug: Trans-resveratrol extract from Polygonum Cuspidatum
- Placebo (Placebo Comparator): All subjects underwent a 2-week run-in period during which placebo was administered. The placebo was manufactured so that it was not distinguishable by color, form, or taste from the active drug. Following the run-in period, subjects who were tolerant of the placebo would proceed to the treatment period. Subjects were given a starting dose of 500 mg daily of matching placebo and instructed to abstain from foods with high resveratrol content during the entire duration of the trial. The dose was increased by 500 mg per day every 3 days to a maximum dose of 3 g per day in three divided doses if there was no hypoglycemia.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trans-resveratrol extract from Polygonum Cuspidatum — Starting dose of 500 mg daily of either resveratrol to be administered on Day 1 and increased by 500 mg per day every 3 days to a maximum dose of 3 g per day in three divided doses if there was no hypoglycemia.
  Other Names: Mega Resveratrol, Danbury, USA
  Arms: Resveratrol
Drug: Placebo
  Arms: Placebo

SUMMARY:
Animal studies indicate that resveratrol, a phytoalexin enriched in the skin of red grapes and a constituent of red wine, is associated with longevity likely through the increased production of a protein, SIRT1.

The trial is a proof-of-concept study primarily designed to examine for the first time in humans, the effect of 12 weeks of oral resveratrol on skeletal muscle SIRT1 expression in 10 patients with T2DM in a randomized, placebo-controlled, double-blind fashion. Secondary outcomes include measures of AMPK, p-AMPK and GLUT4 expression levels, energy expenditure, physical activity levels, distribution of abdominal adipose tissue and skeletal muscle fiber type composition, body weight, HbA1c, plasma lipid subfraction, adiponectin levels and insulin sensitivity.

DETAILED DESCRIPTION:
Eligible criteria include Chinese males, aged between 40 and 69 years old, with T2DM with a HbA1c of 7.1 to 12% and who have been on a stable oral hypoglycemic regimen for the past 3 months. Subjects who were insulin-dependent, with renal or liver impairment or who were terminally ill were excluded.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent
2. Chinese Male
3. Age 40 to 69 yrs old
4. For subjects with type 2 diabetes mellitus

   * Diagnosis of type 2 diabetes mellitus based on MOH criteria and,
   * HbA1c >6.5 during screening

Exclusion Criteria:

Willing to abstain from ingesting large quantities of resveratrol-containing foods (eg. red wine, nuts) Cancer diagnosis that is currently under treatment, is clinically detectable, or that has been treated within the past 5 years Terminal disease or on palliative care Current excessive alcohol intake (>21 units per week for men; 14 units per week for women) On maximal doses of 3 or > oral hypoglycaemic agents On insulin therapy or known type 1 diabetes mellitus Past history of documented or suspected hypoglycemia within last 3 months Past history of recurrent hypoglycemia Past history of serious hypoglycemia as defined by documented hypoglycemia requiring hospital admission Past history of hyperglycemic emergencies within last 6 months Past or current history of hemorrhagic strokes On anti-platelet agents, non-steroidal anti-inflammatory drugs (NSAIDs), anti-coagulation therapy or omega-3 fatty acids History of unexplained bleeding disorders History of any grape allergy History of allergy to local anaesthetic History of surgery with surgery with clips, staples or stents Presence of cardiac pacemaker or metallic foreign body in any part of the body On alternative or traditional medications Treated with another investigational drug within last 6 months Poorly controlled hypertension (SBP >/= 160 or DBP >/= 100) within last one month ALT and/or AST > 1.5 times above upper limit of normal within last 6 months GFR < 50 ml/min/1.73m2 (MDRD equation) within last 6 months

Ages: 40 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-12; Primary Completion 2010-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle sirtuin 1 (SIRT1) expression | 3 months

SECONDARY OUTCOMES:
Skeletal muscle 5'-AMP-activated protein kinase (AMPK) expression | 3 months
Skeletal muscle phosphorylated-AMPK-Thr172 (p-AMPK) expression | 3 months
Skeletal muscle glucose transporter type 4 (GLUT 4) expression | 3 months
Glycated hemoglobin (HbA1c) | 3 months
Body weight | 3 months
Insulin sensitivity | 3 months
Lipid profile | 3 months
Energy expenditure | 3 months
Physical activity level | 3 months
Abdominal adipose tissue distribution | 3 months
Skeletal muscle fibre type composition | 3 months
Renal function | 3 months
  Serum creatinine
Liver function | 3 months
  Transaminases

CONTACTS AND LOCATIONS:
Overall Officials: Kian Peng Goh, FRCP, Principal Investigator — Alexandra Health, Khoo Teck Puat Hospital
Locations (1):
- Alexandra Health, Khoo Teck Puat Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Baur JA, Pearson KJ, Price NL, Jamieson HA, Lerin C, Kalra A, Prabhu VV, Allard JS, Lopez-Lluch G, Lewis K, Pistell PJ, Poosala S, Becker KG, Boss O, Gwinn D, Wang M, Ramaswamy S, Fishbein KW, Spencer RG, Lakatta EG, Le Couteur D, Shaw RJ, Navas P, Puigserver P, Ingram DK, de Cabo R, Sinclair DA. Resveratrol improves health and survival of mice on a high-calorie diet. Nature. 2006 Nov 16;444(7117):337-42. doi: 10.1038/nature05354. Epub 2006 Nov 1. PMID 17086191
- [Background] Lagouge M, Argmann C, Gerhart-Hines Z, Meziane H, Lerin C, Daussin F, Messadeq N, Milne J, Lambert P, Elliott P, Geny B, Laakso M, Puigserver P, Auwerx J. Resveratrol improves mitochondrial function and protects against metabolic disease by activating SIRT1 and PGC-1alpha. Cell. 2006 Dec 15;127(6):1109-22. doi: 10.1016/j.cell.2006.11.013. Epub 2006 Nov 16. PMID 17112576
- [Background] Baur JA, Sinclair DA. Therapeutic potential of resveratrol: the in vivo evidence. Nat Rev Drug Discov. 2006 Jun;5(6):493-506. doi: 10.1038/nrd2060. Epub 2006 May 26. PMID 16732220
- [Background] Fujii N, Jessen N, Goodyear LJ. AMP-activated protein kinase and the regulation of glucose transport. Am J Physiol Endocrinol Metab. 2006 Nov;291(5):E867-77. doi: 10.1152/ajpendo.00207.2006. Epub 2006 Jul 5. PMID 16822958